CLINICAL TRIAL: NCT06749275
Title: Non-invasive Treatment for Root Caries Lesions in Older Adults with Cognitive Impairment
Brief Title: High Fluoride and Root Caries in Older Adults (NIT-RCL-UTALCA)
Acronym: SDF-RCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Responsible Party: Principal Investigator, Soraya León Araya, Associate Professor, University of Talca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDF-RCL-SLeón
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Root Caries; Cognitive Impairment; Fluor
MeSH Terms: conditions — Root Caries; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The total sample (132 individuals) will be divided randomly into 3 groups (44 per group) by means of a listing and using the online software http://www.random.org/ following a simple 1: 1: 1 assignment procedure in each group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Fluoridated products and the different concentrations of toothpastes will be camouflaged and labeled by a member of the research team that does not participate in the clinical study who will keep them in separate boxes prior to delivery. The principal investigator and the outcomes assessor will not know the treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5,000 ppm fluoride toothpaste (Active Comparator): Toothbrushing twice per day with 5,000 ppm fluoride toothpaste + individualized Oral Hygiene Instruction (OHI).
  Toothpaste of 5,000 ppm of fluoride are considered as the control, since according to international clinical guidelines (Slayton et al. 2018) it would be the treatment of choice to treat RCLs.
  Interventions: Device: 5,000 ppm fluoride toothpaste
- 22,600 ppm fluoride varnish (Experimental): Applications of 5% fluoride varnish (22,600 ppm) every 3 months + toothbrushing twice per day with 1,450 ppm fluoride toothpaste + individualized OHI.
  Interventions: Device: 22,600 ppm fluoride varnish
- 38% SDF (Experimental): Biannual applications of 38% SDF solution + toothbrushing twice per day with 1,450 ppm fluoride toothpaste + individualized OHI.
  Interventions: Device: 38% SDF

INTERVENTIONS:
Device: 5,000 ppm fluoride toothpaste — In group 1, toothbrushing with toothpaste of 5,000 ppm of fluoride twice per day for two minutes, after breakfast and before bedtime. Participants will be also instructed not to rinse with water after brushing and to only eliminate the excess of the dentifrice by spitting out. The amount of toothpaste to be used had to be about the size of a pea.
  Other Names: Caristop 5,000 ppm
  Arms: 5,000 ppm fluoride toothpaste
Device: 22,600 ppm fluoride varnish — The application protocol of 5% fluoride varnish will be used together with the 1,450 ppm paste with the same protocol of the group 1: toothbrushing with toothpaste of 1.450 ppm of fluoride twice per day for two minutes, after breakfast and before bedtime. Participants will be also instructed not to rinse with water after brushing and to only eliminate the excess of the dentifrice by spitting out. The amount of toothpaste to be used had to be about the size of a pea.
  Other Names: Duraphat 22.600 ppm
  Arms: 22,600 ppm fluoride varnish
Device: 38% SDF — The application protocol of 38% SDF annually will be used together with the 1,450 ppm paste with the same protocol of the group 2: toothbrushing with toothpaste of 1.450 ppm of fluoride twice per day for two minutes, after breakfast and before bedtime. Participants will be also instructed not to rinse with water after brushing and to only eliminate the excess of the dentifrice by spitting out. The amount of toothpaste to be used had to be about the size of a pea.
  Other Names: Fagamin 44,800 ppm
  Arms: 38% SDF

SUMMARY:
This project aims to provide an effective solution for root caries lesions (RCLs), specifically in older persons with cognitive impairment through a non-invasive therapy with Silver Diamine Fluoride (SDF). We hypothesize that, due to its remineralizing potential and the cariostatic effect conferred by silver, 38% SDF (biannually applied) will be more effective than 5,000 ppm fluoride toothpastes or 22,600 ppm fluoride varnish in preventing and arresting RCLs in older adults with cognitive impairment. The aim of this project, therefore, is to compare the effectiveness of 38% SDF with high-fluoride toothpaste of 5,000 ppm and 5% fluoride varnish of 22,600 ppm, on the incidence and inactivation of RCLs in older adults with mild cognitive impairment.

A double-blind randomized controlled clinical trial (RCT) will be conducted. One hundred thirty-two 65-year-old or older participants diagnosed as having mild cognitive impairment will be invited to participate. To be eligible, subjects must have at least 5 teeth and 1 active RCLs. Participating older adults with moderate or severe cognitive impairment, dementia, severe dependency, terminal illness, aggressive behavior and alcoholism, will be excluded from the study. Included subjects will be randomly assigned to one of the 3 following study arms (n=44 per group):

* Group 1 (Control): Toothbrushing twice per day with 5,000 ppm fluoride toothpaste
* Group 2: Applications of 5% fluoride varnish (22,600 ppm) every 3 months + toothbrushing twice per day with 1,450 ppm fluoride toothpaste.
* Group 3: Biannual applications of 38% SDF solution + toothbrushing twice per day with 1,450 ppm fluoride toothpaste.

Incidence and lesion inactivation (arrest) using Nyvad's criteria for RCLs will be the primary outcomes to assess the effectiveness of the treatments. Clinical assessment every 6 months up to 2 years will be carried out. RCL incidence and Relative Risk (RR) will be obtained and compared among the treatment groups.

This project will contribute novel scientific evidence on the effectiveness of SDF as a non-invasive therapy for RCLs with special focus on the increasing elderly population with cognitive impairment. The results of this project can be readily translated into dental practice to provide an effective and low-cost non-invasive tool to treat RCLs in cognitive impaired population, with potential implications in public health.

DETAILED DESCRIPTION:
This project aims to provide an effective solution for RCLs, specifically in older persons with cognitive impairment through a non-invasive therapy with SDF. SDF has a cariostatic effect - unlike any other fluoridated product -, does not require patient compliance, only needs one annual or biannual application, is easy to manipulate even at home care and is a low-cost product. Root caries is a highly prevalent oral health problem in the elderly population, and it is estimated to increase significantly over time, particularly in people with cognitive impairment. Therapies intended for RCLs have been mostly restorative and highly heterogeneous. Furthermore, clinical management of RCLs, especially in subjects with cognitive impairment, is challenging for the clinician. Limited evidence supports the non-invasive treatment of RCLs, some of them with SDF. In people with cognitive impairment, however, no evidence has been reported, but this approach could be the most advantageous for this complex population. Thus, SDF for RCLs management in this population appears as a novel and attractive solution to the problem. The present study corresponds to a blind randomized controlled clinical trial (RCT) according to the CONSORT (Consolidated Statement of Reporting Trials) statement (Moher et al. 2012), with 3 parallel groups. The total sample (132 individuals) will be divided randomly into 3 groups (44 per group) by means of a listing and using the online software http://www.random.org/ following a simple 1: 1: 1 assignment procedure in each group, prepared by a researcher without clinical participation in the RCT, in order to keep clinical researchers blind. This person will also be responsible for recruiting patients and assigning them to the appropriate group.

The participants of this study will belong to a day center located in Talca, Chile, focused in providing care to people over 65 years of age or older, with cognitive impairment.

Sample size: The sample size was determined for the ANOVA test of repeated measurements using G* Power. The a priori analysis considered an average effect size (ie, 0.3), a 5% error, a statistical power of 80% and a correlation between the initial and final measurements of 0.8, considering a 30% loss rate, according to a previous study (Tan et al. 2010). This calculation gives a total sample of 132 individuals, which would correspond to 44 participants per group.

Intervention and clinical examination: Participants will be randomly assigned to one of the three treatment groups:

• Group 1 or Control: Toothbrushing twice per day with 5,000 ppm fluoride toothpaste + individualized Oral Hygiene Instruction (OHI).

Toothpaste of 5,000 ppm of fluoride are considered as the control, since according to national (MINSAL 2015) and international clinical guidelines (Slayton et al. 2018) it would be the treatment of choice to treat RCLs, when there is strict compliance. Toothbrushing twice per day for two minutes, after breakfast and before bedtime. To increase F concentration and retention, participants will be also instructed not to rinse with water after brushing and to only eliminate the excess of the dentifrice by spitting out. The amount of toothpaste to be used had to be about the size of a pea. This protocol is based on previous studies (León et al. 2019).

• Group 2: Applications of 5% fluoride varnish (22,600 ppm) every 3 months + toothbrushing twice per day with 1,450 ppm fluoride toothpaste + individualized OHI.

The indication for the use of 1,450 ppm fluoride toothpaste is according to the same protocol indicated above (León et al. 2019), for group 2 and 3. In the case of group 2, the application protocol of 5% fluoride varnish will be used every 3 months, as recommended by experts for vulnerable older population (Gluzman et al. 2013).

• Group 3: Biannual applications of 38% SDF solution + toothbrushing twice per day with 1,450 ppm fluoride toothpaste + individualized OHI.

The biannual application of the 38% SDF will be on all exposed root surfaces with RCLs. The teeth to be treated will be relatively isolated with cotton rolls or gauze, the surface to be treated will be dried with air and the SDF will be applied with a microbrush for 1 minute and then rinsed with water (Horst et al. 2017).

For the three groups the IHO will be individualized for each case, that is, according to the motor conditions of the patient or caregiver, or the conditions of oral access of the patient, basically focusing on an effective manual brushing according to previous studies (León et al. 2019; Tan et al. 2010).

Each participant will be evaluated at the center, where there will have access to fluoridated drinking water and a comfortable place, with good lighting (natural light and LED headlight) to make the initial diagnosis through an oral exam, where the RCLs will be registered. In addition, the team of researchers will have a portable dental equipment to facilitate the use of triple syringe with air and water, plus the use of ejector which will facilitate the intervention to the group with SDF. Prior to diagnosis, along with the participant and caregiver, the Comprehensive Oral Geriatric Assessment (COGA or VOGI in Spanish) form will be filled out, containing 4 items (Annex 1): sociodemographic information, systemic condition, oral health history and oral health exam. The filling time by the researcher of the COGA file, plus the total duration of the procedure, should not exceed 30 minutes. In cases where there is accumulation of bacterial plaque or calculus that makes clinical evaluation difficult, a previous supragingival scaling with or without root planning will be performed with manual instruments (curettes and jackets) and subsequently the diagnosis of RCLs will be made.

Fluoridated products and the different concentrations of toothpastes will be camouflaged and labeled by a member of the research team that does not participate in the clinical study who will keep them in separate boxes prior to delivery. The follow-up and evaluation of the outcomes will be carried out at the baseline and after 2 years. Oral and written instructions about the protocol for treatment with toothpastes will be given to participants and their caregivers. Additional toothbrushes and toothpastes will be provided to the volunteers every three months and adherence to treatment will be checked by returning the used dentifrices and toothbrushes to the investigators.

ELIGIBILITY:
Inclusion Criteria:

* People 65 years of age or older, with regular attendance at the Amancay day center at least once a week or belonging to the subsample with mild cognitive impairment of the MAUCO cohort.
* Medical diagnosis of mild cognitive impairment previously made by the psychiatrist of the Amancay team or by the MAUCO study and based on the diagnostic criteria of the International Association of Psychogeriatrics (Levy 1994).
* Have at least 5 teeth in the mouth and 1 active RCLs, according to the methodology of previous studies (León et al. 2019; Tan et al. 2010).
* To be able to do the toothbrushing yourself or, if you cannot do it, allow the person in charge to do it.

Exclusion Criteria:

* Severe dependent older adults and terminal patients (determined according to information from the Amancay team or by the MAUCO study).
* Aggressive older adults (who present aggressive or risky attitudes towards a member of the research team during visits).
* Alcoholic older adults (determined according to information from the Amancay team or by the MAUCO study).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 179 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Root caries | at 6, 12, 18 and 24 months
  Activity status of root caries lesions will be clinically assessed

CONTACTS AND LOCATIONS:
Overall Officials: Soraya León Araya, PhD, Principal Investigator — University of Talca
Locations (1):
- Faculty of Dentistry, Talca, Maule Region, Chile